CLINICAL TRIAL: NCT06327334
Title: Brain Heart InterActioNs in Cardiac Arrest. Ancillary Study of the HEAVENwARd Trial
Acronym: BHIANCA
Status: Recruiting | Type: Observational
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/03
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Arrest
Keywords: Brain-heart interactions; Resuscitated cardiac arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Despite advances in post-resuscitation care of patients with cardiac arrest (CA), the majority of survivors who are treated after restoration of spontaneous circulation (ROSC) will have sequelae of hypoxic-ischemic brain injury ranging from mild cognitive impairment to a vegetative state. Current recommendations suggest using a multimodal approach to predict poor prognosis, meaning combining markers together. Yet, a substantial proportion of patients do not have a clear prognostic evaluation even when applying the latest ESICM recommendations algorithm published in 2021. It is therefore important to identify new prognostic markers to predict both unfavorable and favorable outcomes. Data regarding the pathophysiological mechanisms of post-anoxic encephalopathy suggest a diffuse anoxo-ischemic injury. However, post-mortem neuropathology data suggest that these lesions do not uniformly affect neuroanatomical structures, with some regions (especially hippocampal and insular) appearing more sensitive to anoxia. Conversely, the brainstem appears less affected by anoxic lesions. Under physiological conditions, there are interactions between the heart and the brain, and between the brain and the heart mainly related to the autonomic nervous system, through interactions between central cortical control structures (especially insular) and brainstem structures (at the level of the bulb) and peripheral structures of the heart. Exploring the pathophysiological mechanisms of heart-brain interactions post-CA could thus help better understand the pathophysiology of anoxo-ischemic encephalopathy, before considering potential therapeutic targets. Furthermore, this heart-brain dysfunction could have prognostic value. Indeed, recent studies in healthy subjects and patients with consciousness disorders suggest that autonomic nervous system activity measured by brain-heart interactions could be a reliable marker of consciousness and cognitive processing. These coupled heart-brain interactions can be evaluated through synchronous electroencephalogram (EEG) and electrocardiogram (ECG) recordings, as there are coupled interactions between the signals of these two organs. The existence of abnormal brain-heart coupling could be associated, on the one hand, with the severity of post-anoxic encephalopathy, and on the other hand, with neurological prognosis in patients with persistent coma post-CA.

This ancillary study of a multicentre prospective cohort "HEAVENwARd study" (NCT06044922) will assess the prevalence and prognostic value of bilateral brain-heart interactions in comatose patients after CA.

DETAILED DESCRIPTION:
The study BHIANCA will be an ancillary study of the HEAVENwARd study : HEart rAte Variability in Early prediction of a Noxic brain injury after cardiac ARrest (NCT06044922).

All patients included in the HEAVENwARd study who have an EEG with ECG lead recorded for a neuroprognostication are eligible.

ELIGIBILITY:
Inclusion Criteria:

* Admitted in intensive care unit (ICU) after resuscitation from cardiac arrest (in-hospital or out-of-hospital)
* Coma (Glasgow score < 8) after ROSC, requiring sedation and targeted temperature management for at least 24h
* EEG with ECG lead performed in routine care

Exclusion Criteria:

* Dying patient (Limitation of life support techniques at admission to the ICU)
* Limitation of life sustaining treatment before EEG
* Non-Sinus Rhythm
* Pregnant or breastfeeding women
* Patient under protection of the adults (guardianship, curators or safeguard of justice)
* Opposition by the trusted person or by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Comatose patients admitted in ICU after resuscitation from cardiac arrest
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Bilateral brain-heart interactions | At day-28
  Coupling coefficient between the time-varying power of EEG in different frequency bands and heart rate variability metrics reflecting sympathetic and parasympathetic tone will be compared between post-cardiac arrest patients and normal values in healthy subjects (already acquired database coming from Monin et al. Neurophysiologie Clinique 2018).

SECONDARY OUTCOMES:
Poor neurological outcome evaluated using the CPC score | At day-28
  The CPC (Cerebral Performance Category) score assesses neurological status after cardiac arrest on a scale of 1 to 5 (1 = conscious and normal; 2 = conscious with moderate disability; 3 = conscious with severe disability; 4 = coma or vegetative state; 5 = death).
  The CPC score will be dichotomized as follow: good neurological outcome for categories 1 and 2 and poor neurological outcome or death for categories 3, 4 and 5.
  The CPC score will be obtained at day-28 from an in-hospital visit if the patient is still hospitalized or by phone call if patient returned home.
Mortality | At day-28
Post-anoxic encephalopathy severity evaluated by composite prognostic markers combining EEG patterns, somatosensory evoked potentials (SEP) and neuron specific enolase (NSE). | At day-28

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Brest University Hospital, Brest, Brittany Region
  - Nantes University Hospital, Nantes, Pays de la Loire Region
  - Marseille University Hospital, Marseille, Provence-Alpes-Côte d'Azur Region
  - Ambroise Paré - Hartmann Private Hospital Group, Neuilly-sur-Seine, Île-de-France Region
  - Cochin Hospital, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No